CLINICAL TRIAL: NCT01587274
Title: A Randomized Three-armed Comparative Effectiveness Study of Various Medications for Musculoskeletal Low Back Pain: Defining the Added Benefit of Muscle Relaxants and Opioids.
Brief Title: A Randomized Study of Three Medication Regimens for Acute Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Associate professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-10-379
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Acute Low Back Pain
Keywords: low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Naproxen; cyclobenzaprine; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Opioid (Active Comparator): Naproxen + opioid
  Interventions: Drug: Naproxen; Drug: Oxycodone/ acetaminophen
- Skeletal muscle relaxant (Active Comparator): Naproxen + skeletal muscle relaxant
  Interventions: Drug: Naproxen; Drug: Cyclobenzaprine
- Naproxen alone (Active Comparator): Naproxen + placebo
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: Naproxen — Naproxen 500mg twice/ day x 10 days
Drug: Cyclobenzaprine — Cyclobenzaprine 5-10mg three times/ day x 10 days
  Arms: Skeletal muscle relaxant
Drug: Oxycodone/ acetaminophen — Oxycodone 5-10mg/ Acetaminophen 325-650 mg three times/ day x 10 days
  Arms: Opioid

SUMMARY:
Low back pain causes 2.4% of visits to US emergency departments (ED) resulting in 2.7 million visits annually. In a general low back pain (LBP) population, prognosis is poor. About 50% of patients who visited general practitioners with new onset musculoskeletal LBP report persistent pain and functional disability three months after the index visit. Outcomes are similarly poor for the population of patients forced to use an ED for management of their LBP. In an observational study of patients with non-traumatic LBP recently completed at the PI's institution, patients were contacted one week after ED discharge: 70% reported persistent back-pain related functional impairment, 59% reported moderate or severe LBP, and 69% reported analgesic use within the previous 24 hours. Three months after the ED visit, 48% reported functional impairment, 42% reported moderate or severe pain, and 46% reported analgesic use within the previous 24 hours.

A variety of evidence-based medications are available to treat LBP. Non-steroidal anti-inflammatory drugs (NSAID) are more efficacious than placebo with regard to pain relief, global improvement, and requirement of analgesic medication. Skeletal muscle-relaxants too are effective for short-term pain relief and global efficacy. Opioids are commonly used for moderate or severe acute LBP,(9) though high-quality evidence supporting this practice is lacking.

Treatment of LBP with multiple concurrent medications is common in the ED setting. Emergency physicians often prescribe NSAIDs, skeletal muscle relaxants, and opioids in combination. Several clinical trials have compared combination therapy with NSAIDS+ skeletal muscle relaxants to monotherapy with just one of these agents. These trials have reported heterogeneous results. The combination of opioids + NSAIDS has not been evaluated experimentally in patients with acute LBP.

Given the poor pain and functional outcomes that persist beyond an ED visit for musculoskeletal LBP, the investigators propose a clinical trial to evaluate whether combining muscle relaxants or opioids with NSAIDs is more effective than NSAID monotherapy for the treatment of non-traumatic, non-radicular low back pain. Specifically, the investigators will evaluate three distinct hypotheses:

1. The combination of naproxen + cyclobenzaprine will provide greater relief of LBP than naproxen alone seven days after an ED visit, as measured by the Roland Morris low back pain functional disability scale
2. The combination of naproxen + oxycodone/ acetaminophen will provide greater relief of LBP than naproxen alone seven days after an ED visit, as measured by the Roland Morris low back pain functional disability scale
3. The combination of naproxen + oxycodone/ acetaminophen will provide greater relief of LBP than naproxen + cyclobenzaprine seven days after an ED visit, as measured by the Roland Morris low back pain functional disability scale

ELIGIBILITY:
Inclusion Criteria:

* Non-radicular, non-traumatic low back pain of no more than 2 weeks duration

Exclusion Criteria:

* Back pain longer than 2 weeks
* Prior to the acute attack of low back pain, back pain once per month or more frequently
* Prior to the acute attack of low back pain, daily or near daily use of pain medication

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 323 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Friedman BW, Dym AA, Davitt M, Holden L, Solorzano C, Esses D, Bijur PE, Gallagher EJ. Naproxen With Cyclobenzaprine, Oxycodone/Acetaminophen, or Placebo for Treating Acute Low Back Pain: A Randomized Clinical Trial. JAMA. 2015 Oct 20;314(15):1572-80. doi: 10.1001/jama.2015.13043. PMID 26501533

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Opioid | Skeletal Muscle Relaxant | Naproxen Alone
Started | 108 | 108 | 107
Completed | 104 | 103 | 104
Not Completed | 4 | 5 | 3
Not completed — Lost to Follow-up | 4 | 5 | 3

BASELINE CHARACTERISTICS:
Population: Patients enrolled and randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid | Skeletal Muscle Relaxant | Naproxen Alone | Total
Number analyzed (Participants) | 108 | 108 | 107 | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (11) | 38 (11) | 39 (11) | 39 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 45 | 53 | 158
  Male | 48 | 63 | 54 | 165
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 108 | 108 | 107 | 323
Pre-existing functional impairment as measured by the Roland Morris Disability Questionnaire [Median (Inter-Quartile Range); unit: units on a scale] — The Roland Morris Disability Questionnaire (RMDQ) is a 24 item instrument that evaluates the impact of low back pain on one's daily life. It is most sensitive for patients with mild to moderate disability due to acute, sub-acute or chronic low back pain. Each question can be answered as either a "yes" or "no". The score ranges from 0 to 24 where a higher score reflects greater impairment and, therefore, worsening in the quality of life.
  units on a scale | 20 [17 to 22] | 19 [17 to 21] | 20 [17 to 21] | 20 [17 to 21]

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Disability as Measured by the Roland Morris Disability Questionnaire
Description: The Roland Morris Disability Questionnaire (RMDQ) is a 24 item instrument that evaluates the impact of low back pain on one's daily life. It is most sensitive for patients with mild to moderate disability due to acute, sub-acute or chronic low back pain. Each question can be answered as either a "yes" or "no". The score ranges from 0 to 24 where a higher score reflects greater impairment and, therefore, worsening in the quality of life. The change in RMDQ is obtained by subtracting the RMDQ score at one week after discharge from the baseline score.
Time Frame: Baseline and one week after discharge from emergency department
Population: Multiple imputation used to account for participants lost to follow-up
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Opioid | Skeletal Muscle Relaxant | Naproxen Alone
Number analyzed (Participants) | 108 | 108 | 107
units on a scale | 5 [0 to 15] | 4 [0 to 16] | 7 [0 to 18]

ADVERSE EVENTS:
Arm/Group | Opioid | Skeletal Muscle Relaxant | Naproxen Alone
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/108 | 0/107
Other Adverse Events (participants affected / at risk) | 43/108 | 36/108 | 22/107
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Opioid (N=108) | Skeletal Muscle Relaxant (N=108) | Naproxen Alone (N=107)
Nausea/ vomiting (Gastrointestinal disorders) | 19 | 4 | 6
Drowsiness (Nervous system disorders) | 16 | 7 | 4
Dizziness (Nervous system disorders) | 16 | 7 | 4
Stomach irritation (Gastrointestinal disorders) | 7 | 7 | 5
Other (Investigations) | 0 | 11 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes